CLINICAL TRIAL: NCT07006077
Title: A Phase II Trial to Evaluate the Efficacy of Recombinant Human IL-21-expressing Oncolytic Vaccinia Virus Injection (hV01) in Patients With Advanced Pancreatic Tumors
Brief Title: Recombinant Human IL-21-expressing Oncolytic Vaccinia Virus Injection (hV01) in Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Converd Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hV01-ITu-202
Record Dates: First submitted 2025-05-09; First posted 2025-06-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Advanced Pancreatic Cancer
Keywords: phase Ⅱ; vaccinia virus; IL-21; Pancreatic Tumors
MeSH Terms: conditions — Vaccinia; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hV01 intratumoral injection (Experimental): Participants will receive intratumoral injections of hV01 at the dose level of 8.0×10^8 PFU on Day 1 and Day 15 of each treatment cycle.
  Interventions: Biological: Recombinant human IL-21-expressing oncolytic vaccinia virus injection

INTERVENTIONS:
Biological: Recombinant human IL-21-expressing oncolytic vaccinia virus injection — hV01 is a recombinant vaccinia virus with deletions of the viral thymidine kinase (TK) and viral growth factor (VGF) genes and insertion of the human IL-21 gene.

SUMMARY:
The main goal of this clinical trial is to preliminary evaluate the efficacy of recombinant human IL-21-expressing oncolytic vaccinia virus injection (hV01) in patients with advanced pancreatic cancer.And the secondary purpose is to evaluate the safety of hV01.

DETAILED DESCRIPTION:
This is a single-site, single-arm, open-label,exploratory phase Ⅱa study. Based on the safety results of the completed phase I clinical trial of hV01 , 8.0x10 ^ 8 PFU was selected as a dose level of the dosage for each administration in this clinical trial, hV01 will be administered with twice per cycle (on day 1 and day 15), efficacy evaluation will be conducted on day 28, and every 28 days as a treatment cycle,during which safety will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Signing an informed consent form.
* Men or women aged 18 to 75 years.
* Histologically and/or cytologically confirmed advanced malignant advanced pancreatic tumors refractory or failed to respond to standard therapy (including disease progression and/or intolerable toxicities).
* At least one measurable lesion according to RECIST v1.1 criteria, which can be injected intratumorally either directly or with the assistance of Endoscopic ultrasound. The baseline longest diameter (shortest diameter for lymph node lesions) of the lesion targeted for injection should be more than 1.5 cm, and the lesion also meets the requirements of the relevant dosing volume.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Required baseline laboratory data include:

  a) Hematology: absolute neutrophil count (ANC) ≥ 1.5×10^9/L, platelet (PLT) count ≥ 75×10^9/L, hemoglobin (Hb) ≥90 g/L (without supportive therapy within 14 days prior to laboratory test); b) Liver function: serum total bilirubin (TBIL) ≤1.5×ULN (or ≤3×ULN for patients with liver metastasis); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN (or<5×ULN for patients with primary liver cancer or liver metastasis); c) Renal function: serum creatinine (Cr) ≤1.5×ULN, and creatinine clearance (Cockcroft-Gault method) ≥45 mL/min. For men: creatinine clearance = [[140-age(yr)]×weight (kg)]/[0.818×creatinine (μmol/L)]; For women: creatinine clearance = [[140-age(yr)]×weight (kg)×0.85]/[0.818×creatinine (μmol/L)]; d) Coagulation test: activated partial thromboplastin time (APTT) ≤1.5×ULN; international normalized ratio (INR) ≤1.5×ULN.
* Female patients of childbearing age must have a negative serum pregnancy test. Female patients of childbearing age and male patients whose partners are of childbearing age must agree to use medically approved contraceptive measures (hormonal or barrier methods or abstinence) throughout the treatment period and also within 3 months after the last dose of the investigational drug. Male patients must also avoid sperm donation.

Exclusion Criteria:

* Receiving any of the following anti-tumor treatments within a specified time period:

  a) Systemic anti-tumor treatment, including chemotherapy, large-molecule targeted therapy, immunotherapy, and endocrine therapy within 4 weeks before first dose (within 6 weeks of dosing for nitrosourea or mitomycin C); b) Small-molecule targeted therapy within 2 weeks before first dose or within 5 half-lives of the small-molecule targeted drug (whichever is longer); c) Traditional Chinese medicine or Chinese herbal medicine used as anti-tumor agent within 2 weeks before first dose; d) Radiotherapy (excluding palliative radiotherapy) within 2 weeks before first dose; e) Prior oncolytic virus treatment.
* Acute toxic effects from prior treatments not resolved to Common Terminology Criteria for Adverse Events (CTCAE, v5.0) grade 1 or below, except for toxicities deemed safe by the investigator, such as alopecia.
* Patients with clinical symptoms of central nervous system (CNS) metastasis or meningeal metastasis, or other evidence indicating that CNS or meningeal metastases are not controlled.
* Known or suspected active autoimmune diseases (including but not limited to systemic lupus erythematosus, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, and Hashimoto's thyroiditis).
* History of severe cardiovascular and cerebrovascular diseases, including:

  a) Acute coronary syndrome (including myocardial infarction, severe or unstable angina), myocarditis, congestive heart failure, cerebrovascular accidents, or other cardiovascular events of CTCAE (v5.0) grade 3 or higher within 12 months of dosing; b) Severe arrhythmia requiring clinical intervention (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes), corrected QT interval (QTc) >450 ms for males or >470 ms for females, or a family history of long QT syndrome; c) New York Heart Association (NYHA) classification of class II or above, or left ventricular ejection fraction (LVEF) <50%; d) Uncontrolled hypertension (as judged by the investigator) or hypotension despite standard treatment.
* Any uncontrolled active infection requiring systemic anti-infective therapy (graded 2 or higher according to CTCAE v5.0), including but not limited to active tuberculosis, sepsis, bacteremia, fungemia, and viremia.
* Any of the following infections: human immunodeficiency virus (HIV), syphilis spirochete(TP), active hepatitis C (positive HCV RNA test) or active hepatitis B (positive HBsAg and HBV DNA ≥ 2000 IU/mL or ≥10^4 copies/mL).
* Use of immunomodulatory drugs within 2 weeks of dosing, including but not limited to thymosin, interleukin, interferon.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Anti-tumor activity of hV01: overall response rate (ORR). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the overall response rate (ORR) as a measurement of tumor response and disease progression.
Anti-tumor activity of hV01: disease control rate (DCR). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the disease control rate (DCR) as a measurement of tumor response and disease progression.
Anti-tumor activity of hV01: duration of response (DOR). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the duration of response (DOR) as a measurement of tumor response and disease progression.

SECONDARY OUTCOMES:
Anti-tumor activity of hV01: progression-free survival (PFS). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the progression-free survival (PFS) as a measurement of tumor response and disease progression.
Preliminary efficacy of hV01: overall survival (OS). | From signing informed consent form until the date of death from any cause, assessed up to 2 years after the end of treatment.
  To evaluate the overall survival (OS) as a measurement of preliminary efficacy.
To assess the adverse events (AEs) and tolerability of hV01. | From informed consent till 28 days after first dose.
  To assess the frequency, severity, and nature of adverse events (AEs) of hV01 administered by multiple intratumoral injections by a predetermined dose levels of 8x10^8 PFU. This will be determined by abnormalities or changes in vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, 12-lead electrocardiogram, and laboratory test results.

OTHER OUTCOMES:
morphological assessment of tumor cells | Day 1 and Day 15 of every treatment cycle，From baseline until the End of Treatment
  To compare the morphological characteristics of tumor cells before and after administration
To assess immune cells in the peripheral blood | From baseline to 4 weeks after the End of Treatment.
  To assess the levels of lymphocytes (CD3+ cells, CD3+CD4+ cells, CD3+CD8+ cells, CD3+CD4+/CD3+CD8+, CD3-CD16+CD56+ cells, CD3-CD19+ cells) in the peripheral blood.
To assess the expression levels of TILs and protein markers in tumor tissue. | Day 1 and Day 15 of every treatment cycle，From baseline until the End of Treatment
  To assess the expression levels of infiltrating lymphocytes (TILs) and protein markers such as PD-L1, HER2, CTLA-4 in tumor tissue before and after hV01 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, Principal Investigator — Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University
Locations (1):
- Affiliated Hangzhou First People's Hospital,School of Medicine,Westlake University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No